CLINICAL TRIAL: NCT00884403
Title: Gestational Age is Underestimated by Menstrual Dating Compared to Ultrasound Dating in Those Undergoing Abortion up to 20 Weeks
Status: Terminated | Type: Observational
Why Stopped: This study is a retrospective chart review study, not a clinical trial.
Sponsor: University of British Columbia (Other)
Collaborators: Women's Health Research Institute of British Columbia (Other)
Responsible Party: Principal Investigator, Wendy Norman, Principle Investigator, University of British Columbia
Other Study IDs: H08-01332
Record Dates: First submitted 2009-04-03; First posted 2009-04-20 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Abortion
Keywords: abortion; pregnancy dating; gestational age; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Several large trials report gestational dating by last menstrual period (LMP) overestimates gestational age (GA) vs. ultrasound (US) by approximately one week. Previous studies examined only term pregnancies. The investigators hypothesize an opposite tendency in women seeking abortion. This is an observational study undertaken by chart review.

DETAILED DESCRIPTION:
Retrospective cohort study by chart review. We propose to review the charts of four thousand women obtaining abortion in British Columbia, BC. Data will be extracted from the charts of women who obtained abortions between January first 2002 and June 30, 2008 inclusive at two abortion clinics in Vancouver, British Columbia: BC Women's Hospital CARE program, and the Elizabeth Bagshaw Women's Clinic. Specifically we will record age, parity, date of LMP, presence of regular cycles, ultrasound estimation of gestational age, ultrasound measurements: crown rump length, bi-parietal diameter, gestational sac diameter if available, date of abortion, estimation of gestational age by examination of the products of conception, and fetal foot length if available. Further we will record associated factors such as contraception at time of conception, intravenous drug use, and regularity of menstrual cycle. We will calculate the gestational age at time of abortion by the LMP date, by the ultrasound date reported, ultrasound date based on the Hadlock protocol by the reported CRL and similarly BPD as well as calculating the gestational age based on the recorded fetal foot length.

ELIGIBILITY:
Inclusion Criteria:

* Included charts of women who obtained abortion up to twenty weeks gestational age must have a stated LMP date, a pre-operative ultrasound, a viable pregnancy at the time of the abortion and an assessment of the gestational age of the products of conception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women in British Columbia who obtained abortion up to twenty weeks gestational age.
Sampling Method: Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Difference between actual gestational age assessed by pre-operative ultrasound and gestational age estimated by menstrual dating | 1 year

SECONDARY OUTCOMES:
Correlation of the difference between AGA and LMP dating with demographic and obstetrical history factors. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wendy V. Norman, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital CARE Program, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Norman WV, Bergunder J, Eccles L. Accuracy of gestational age estimated by menstrual dating in women seeking abortion beyond nine weeks. J Obstet Gynaecol Can. 2011 Mar;33(3):252-7. doi: 10.1016/s1701-2163(16)34826-5. PMID 21453565